CLINICAL TRIAL: NCT01300091
Title: Burden and Outcome of Shoulder Disorders in Primary Health Care
Status: Withdrawn | Type: Observational
Why Stopped: Recruitment not started
Sponsor: Central Finland Hospital District (Other)
Responsible Party: Ilkka Kiviranta, Department of Orthopaedics and Traumatology, Helsinki University Hospital, Helsinki, Finland
Other Study IDs: B07103-3
Record Dates: First submitted 2011-02-18; First posted 2011-02-21 (Estimated); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Shoulder Pain; Shoulder Mobility Impairment
Keywords: Shoulder; Pain; Range of Motion; Disability Evaluation; Function; Sick Leave; Primary Health Care; Visual Analog Scale; Visual Analog Pain Scale; The American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form
MeSH Terms: conditions — Shoulder Pain; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Consumption of medical care and outcome of shoulder pain and disability in primary care.

DETAILED DESCRIPTION:
Shoulder pain and impairment are common in primary health care. The prognosis of several individuals consulting for a new episode of shoulder problem is surprisingly poor. The objectives are to characterize the consumption of medical care and outcome of shoulder pain and disability in primary health care.

A composite questionnaire consisting of demographic information and ASES questionnaire was used to measure the shoulder function. The patients were sent a second questionnaire after one year.

ELIGIBILITY:
Inclusion Criteria:

* All individuals suffering from shoulder pain or impairment

Exclusion Criteria:

* No

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients consulting a general practitioner due to shoulder disorder during the recruitment period are included. The study population consists of two public health centres with a population of 120 000 individuals and two occupational medicine clinics with a population of 15 000 individuals. The population of health centres and occupational health clinics overlap partially.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Consumption of medical care | one year
  Number of consultations, referrals, and radiologic examinations; Use of pain medication; Number of days on sick leave; Number of visits to physiotherapist; Number of surgical procedures

SECONDARY OUTCOMES:
Development of the ASES score | one year
  ASES score: the patient self-report section of the American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form

CONTACTS AND LOCATIONS:
Locations (1):
- Central Finland Hospital District, Jyväskylä, Finland

REFERENCES:
- [Background] Dorrestijn O, Greving K, van der Veen WJ, van der Meer K, Diercks RL, Winters JC, Stevens M. Patients with shoulder complaints in general practice: consumption of medical care. Rheumatology (Oxford). 2011 Feb;50(2):389-95. doi: 10.1093/rheumatology/keq333. Epub 2010 Nov 2. PMID 21047806
- [Background] Reilingh ML, Kuijpers T, Tanja-Harfterkamp AM, van der Windt DA. Course and prognosis of shoulder symptoms in general practice. Rheumatology (Oxford). 2008 May;47(5):724-30. doi: 10.1093/rheumatology/ken044. Epub 2008 Apr 14. PMID 18411219